CLINICAL TRIAL: NCT04192630
Title: A Study to Document the Safety and Effectiveness of a New Cohesive OVD When Compared to a Control OVD
Brief Title: A Study of B + L Ophthalmic Viscosurgical Device (OVD) CVisc50
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bausch & Lomb Incorporated (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 878
Record Dates: First submitted 2019-12-06; First posted 2019-12-10 (Actual); Results first posted 2024-05-28 (Actual); Last update posted 2024-05-28 (Actual); Status verified 2022-12

CONDITIONS: Cataract
MeSH Terms: conditions — Cataract | interventions — Cataract Extraction

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (2):
- CVisc50 Ophthalmic Viscosurgical Device (OVD) (Experimental): CVisc50 OVD will be carefully injected into the anterior chamber using standard aseptic technique, during the surgical procedure. The duration of the treatment is anticipated to be approximately 15-20 minutes for the surgical procedure. The OVD may also be used to coat surgical instruments prior to Intraocular Lens (IOL) implantation (for example, the internal surfaces of an IOL inserter are typically filled and/or coated with the OVD to provide lubricity during IOL compression and delivery into the eye). Additional OVD of the same product, may be injected as needed throughout surgery to keep the anterior chamber fully formed and to re-inflate the capsular bag following cataract removal. At the end of the surgical procedure it is recommended that OVD be removed from the eye as completely as practical by thoroughly irrigating and aspirating with a sterile irrigating solution.
  Interventions: Device: CVisc50 OVD; Procedure: Cataract Surgery
- ProVisc OVD (Active Comparator): ProVisc OVD will be carefully injected into the anterior chamber using standard aseptic technique, during the surgical procedure. The duration of the treatment is anticipated to be approximately 15-20 minutes for the surgical procedure. The OVD may also be used to coat surgical instruments prior to IOL implantation (for example, the internal surfaces of an IOL inserter are typically filled and/or coated with the OVD to provide lubricity during IOL compression and delivery into the eye). Additional OVD of the same product, may be injected as needed throughout surgery to keep the anterior chamber fully formed and to re-inflate the capsular bag following cataract removal. At the end of the surgical procedure it is recommended that OVD be removed from the eye as completely as practical by thoroughly irrigating and aspirating with a sterile irrigating solution.
  Interventions: Device: ProVisc OVD; Procedure: Cataract Surgery

INTERVENTIONS:
Device: CVisc50 OVD — Bausch + Lomb CVisc50 Cohesive OVD
  Other Names: Bausch + Lomb CVisc50 Cohesive OVD
  Arms: CVisc50 Ophthalmic Viscosurgical Device (OVD)
Device: ProVisc OVD — ProVisc OVD
  Other Names: Alcon ProVisc® OVD
  Arms: ProVisc OVD
Procedure: Cataract Surgery — Cataract Surgery

SUMMARY:
The objective of the study is to evaluate the safety and effectiveness of the Bausch & Lomb CVisc50 cohesive OVD compared to the Alcon ProVisc® cohesive OVD when used in cataract surgery.

DETAILED DESCRIPTION:
The objective of the study is to evaluate the safety and effectiveness of the Bausch & Lomb CVisc50 cohesive OVD compared to the Alcon ProVisc® cohesive OVD when used in cataract surgery.

ELIGIBILITY:
Inclusion Criteria:

* The participant must be at least 45 years old and have a clinically documented diagnosis of age-related non-complicated cataract that is considered amenable to treatment with standard phacoemulsification cataract extraction and IOL implantation.
* The participant must have the capability to provide written informed consent on the Institutional Review Board (IRB)/Ethics Committee (EC) approved Informed Consent Form (ICF) and provide authorization as appropriate for local privacy regulations.
* The participant must be willing and able to undergo all pre-surgical and surgical procedures and to return for all scheduled follow-up examinations through 90 days following surgery.
* The participant must have clear intraocular media other than the cataract in the operative eye.

Exclusion Criteria:

* The participant has participated in any drug or device clinical investigation within 30 days prior to entry into this study and/or plans to do so during the period of study participation.
* The participant has any corneal pathology (for example; significant scarring, guttata, inflammation, edema, dystrophy, etc.) in the operative eye.
* The participant has anterior segment pathology likely to increase the risk of an adverse outcome for phacoemulsification cataract surgery (for example; pseudoexfoliation syndrome, synechiae, iris atrophy, inadequate dilation, shallow anterior chamber, traumatic cataract, lens subluxation) in the operative eye.
* The participant has any condition which prevents reliable specular microscopy in the operative eye.
* The participant has a congenital ocular anomaly (for example; aniridia, congenital cataract) in the operative eye.
* The participant has a baseline ECD <1500 cells/square millimeter (mm^2) in the operative eye.
* The participant has a grade 4+ nuclear cataract density in the planned operative eye.
* The participant has glaucoma or ocular hypertension (IOP >24 mmHg) in the operative eye.
* The participant has any abnormality which prevents reliable Goldmann applanation tonometry in the operative eye.
* The participant has a known allergy to any of the components of the test or control OVDs.
* The participant is using any topical or systemic medications known to interfere with visual performance or complicate cataract surgery within 30 days of enrollment or during the study.
* The participant is scheduled to undergo other combined intraocular procedures during the cataract/intraocular lens (IOL) implantation surgery in the operative eye. NOTE: A relaxing keratotomy is allowed.
* The participant has diabetic retinopathy, wet age-related macular degeneration or other retinal pathology which might limit postoperative visual acuity (VA) or predispose the participant to postoperative retinal complications in the operative eye.
* The participant's fellow eye is already participating in this study.
* The participant has a history of chronic or recurrent inflammatory eye disease (for example; iritis, scleritis, uveitis, iridocyclitis, rubeosis iridis) in the operative eye.
* The participant has a best corrected distance visual acuity (BCDVA) of logarithm of minimum angle resolution (LogMAR) 1.0 (20/200, 6/60) or worse in the fellow eye.
* The participant has had previous corneal surgery in the planned operative eye.
* The participant has a previous retinal detachment in the operative eye.
* Females of childbearing potential (those who are not surgically sterilized or not postmenopausal for at least 12 months) are excluded from participation in the study if they are currently pregnant; plan to become pregnant during the study; and/or are breast-feeding.

Min Age: 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 390 (Actual)
Dates: Start 2019-11-26 (Actual); Primary Completion 2022-01-31 (Actual); Study Completion 2022-01-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Anya Loncaric, Study Director — B+L
Locations (22):
- United States (22):
  - Bausch Site 017, Chandler, Arizona
  - Bausch Site 001, Phoenix, Arizona
  - Bausch Site 008, Fayetteville, Arkansas
  - Bausch Site 010, Burlingame, California
  - Bausch Site 007, Garden Grove, California
  - Bausch Site 011, Newport Beach, California
  - Bausch Site 012, Northridge, California
  - Bausch Site 013, Rancho Cordova, California
  - Bausch Site 004, Torrance, California
  - Bausch Site 019, Bloomington, Minnesota
  - Bausch Site 020, Kansas City, Missouri
  - Bausch Site 002, St Louis, Missouri
  - Bausch Site 015, Washington, Missouri
  - Bausch Site 005, New York, New York
  - Bausch Site 021, Mason, Ohio
  - Bausch Site 003, Reading, Pennsylvania
  - Bausch Site 014, Goodlettsville, Tennessee
  - Bausch 018, Nashville, Tennessee
  - Bausch Site 009, Cedar Park, Texas
  - Bausch Site 006, Houston, Texas
  - Bausch 022, San Antonio, Texas
  - Bausch Site 016, San Antonio, Texas

REFERENCES:
- [Derived] Packer M, Shultz M, Loden J, Lau G. Safety and effectiveness comparison of a new cohesive ophthalmic viscosurgical device. J Cataract Refract Surg. 2023 Aug 1;49(8):804-811. doi: 10.1097/j.jcrs.0000000000001201. PMID 37079390

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | CVisc50 Ophthalmic Viscosurgical Device (OVD) | ProVisc OVD
Started | 194 | 196
Completed | 187 | 193
Not Completed | 7 | 3
Not completed — Discontinued before surgery | 2 | 0
Not completed — Discontinued after surgery | 5 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | CVisc50 Ophthalmic Viscosurgical Device (OVD) | ProVisc OVD | Total
Number analyzed (Participants) | 192 | 196 | 388
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 59 | 65 | 124
  >=65 years | 133 | 131 | 264
Age, Continuous [Mean (Standard Deviation); unit: Years] | 68.7 (7.78) | 67.9 (8.24) | 68.3 (8.01)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 115 | 127 | 242
  Male | 77 | 69 | 146
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 33 | 21 | 54
  Not Hispanic or Latino | 159 | 175 | 334
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 26 | 26 | 52
  Native Hawaiian or Other Pacific Islander | 1 | 2 | 3
  Black or African American | 11 | 19 | 30
  White | 154 | 149 | 303
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 192 | 196 | 388

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Who Experienced at Least One Intraocular Pressure (IOP) Measurement ≥30 Millimeters of Mercury (mmHg) at Any Post-Surgical Follow-up Visit
Time Frame: Up to 90 Days ± 14 Days
Measure: Count of Participants; unit: Participants
Arm/Group | CVisc50 Ophthalmic Viscosurgical Device (OVD) | ProVisc OVD
Number analyzed (Participants) | 192 | 196
Participants | 10 | 16

2. Primary Outcome: Change From Baseline in Corneal Endothelial Cell Density (ECD) in the Study Eye at Postoperative Visit 5 (90 Days ± 14 Days)
Time Frame: Baseline, 90 Days ± 14 Days
Measure: Mean (Standard Deviation); unit: cells/mm2
Arm/Group | CVisc50 Ophthalmic Viscosurgical Device (OVD) | ProVisc OVD
Number analyzed (Participants) | 191 | 195
cells/mm2 | 15.7 (2.80) | 15.8 (3.04)

3. Secondary Outcome: Mean Change From Baseline in IOP at the 6-Hour Post-Operative Visit
Time Frame: Baseline, 6-hour post-operative
Measure: Mean (Standard Deviation); unit: mmhg
Arm/Group | CVisc50 Ophthalmic Viscosurgical Device (OVD) | ProVisc OVD
Number analyzed (Participants) | 191 | 196
mmhg
  Observed value at baseline. | 19.5 (6.53) | 20.0 (6.75)
  Change from baseline. | 3.8 (6.29) | 4.2 (6.87)

4. Secondary Outcome: Mean Change From Baseline in IOP at the 24-Hour Post-Operative Visit
Time Frame: Baseline, 24-hour post-operative
Measure: Mean (Standard Deviation); unit: mmhg
Arm/Group | CVisc50 Ophthalmic Viscosurgical Device (OVD) | ProVisc OVD
Number analyzed (Participants) | 192 | 195
mmhg
  Observed Value at baseline | 18.0 (4.70) | 18.4 (4.78)
  Change from Baseline | 2.3 (4.57) | 2.6 (4.73)

5. Secondary Outcome: Percentage of Participants With Summed Score for Anterior Chamber Cells and Flare Greater Than Zero at the 6-Hour and 24-Hour Post-Operative Visits
Description: Anterior chamber cells were graded on a 6-point scale, with 0 = <1 cell count; 0.5 = 1 to 5 cell count; 1 = 6 to 15 cell count; 2 = 16 to 25 cell count; 3 = 26 to 50 cell count; and 4 = >50 cell count. Anterior chamber flare (protein escaping from dilated vessels) was graded on a 5-point scale, with 0 = none; 1 = faint; 2 = moderate; 3 = marked; and 4 = intense.
Time Frame: 6-hour and 24-hour post-operative
Measure: Count of Participants; unit: Participants
Arm/Group | CVisc50 Ophthalmic Viscosurgical Device (OVD) | ProVisc OVD
Number analyzed (Participants) | 191 | 195
Participants
  6-Hour Post-Operative Visits | 177 | 187
  24-Hour Post-Operative Visits | 183 | 184

ADVERSE EVENTS:
Time Frame: Up to 164 days from preoperative visit to post operative visit 5
Description: Ocular Adverse Event
Arm/Group | CVisc50 Ophthalmic Viscosurgical Device (OVD) | ProVisc OVD
All-Cause Mortality (participants affected / at risk) | 0/192 | 0/196
Serious Adverse Events (participants affected / at risk) | 0/192 | 0/196
Other Adverse Events (participants affected / at risk) | 62/192 | 63/196
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | CVisc50 Ophthalmic Viscosurgical Device (OVD) (N=192) | ProVisc OVD (N=196)
Treatment-Emergent Adverse Events (General disorders) | 62 (75) | 63 (90) — A total of 75 TEAEs were reported for 62 subjects in the CVisc50 group, 90 TEAEs, were reported for 63 subjects in the ProVisc® group. The majority of TEAEs were mild or moderate in both treatment groups

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-08-09): https://cdn.clinicaltrials.gov/large-docs/30/NCT04192630/Prot_SAP_000.pdf